CLINICAL TRIAL: NCT01106131
Title: Efficacy and Safety of CKD-501 or Pioglitazone Added to Ongoing Metformin Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Alone: Multi Center, Randomized, Double Blind, Therapeutic Confirmatory Study
Brief Title: Efficacy and Safety of CKD-501 Versus Pioglitazone When Added to Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19DM09F
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CKD-501 0.5mg (Experimental)
  Interventions: Drug: CKD-501 0.5mg
- Pioglitazone 15mg (Active Comparator)
  Interventions: Drug: Pioglitazone 15mg

INTERVENTIONS:
Drug: CKD-501 0.5mg — CKD-501 0.5mg, orally, 1 tablet once a day for 24weeks or 52weeks(if extension study) with metformin.
  Other Names: Lobeglitazone
  Arms: CKD-501 0.5mg
Drug: Pioglitazone 15mg — Pioglitazone 15mg, orally, 1 tablet or 2 tablet(if confirmed case) once a day for 24weeks with metformin.
  Arms: Pioglitazone 15mg

SUMMARY:
The purpose of this study is to prove effect of glucose reduction that CKD-501 and metformin combination treatment group is non inferiority compare to pioglitazone and metformin combination.

DETAILED DESCRIPTION:
The aim of this phase 3 study was to evaluate the efficacy and safety of CKD-501 and metformin combination for 24 weeks in type 2 diabetes mellitus. Furthermore, the extension study for additional 28weeks is designed to confirm long term safety of CKD-501 as an oral hypoglycemic agent.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 years and 80 years old(male or female)
* Type Ⅱ diabetes mellitus
* The patient who has been taking oral hypoglycemic agent since 2 months with HbA1c 7 to 10% at screening test
* BMI between 21kg/㎡ and 40kg/㎡
* C-peptide level is over 1.0 ng/ml
* Agreement with written informed consent

Exclusion Criteria:

* Type I diabetes or secondary diabetes
* Continuous or non continuous treatment(over 7 days) insulin within 3 month prior to screening
* Treatment with thiazolidinediones within 60 days or patient who have experience such as hypersensitivity reaction, serious adverse event or no effect by treatment with glitazones
* Chronic(continuous over 7 days) oral or non oral corticosteroids treatment within 1 month prior to screening
* Past history: lactic acidosis or metformin contraindication
* Acute or chronic metabolic acidosis including diabetic ketoacidosis
* History of proliferative diabetic retinopathy
* Severe infection, severe injury patients (pre and post operation)
* Oligotrophy,starvation, hyposthenia, pituitary insufficiency or capsular insufficiency
* Drug abuse or history of alcoholism
* History of myocardial infarction, heart failure, cerebral infarction, hematencephalon or unstable angina within 6 months
* Fasting Plasma Glucose level is over 270 mg/dl
* Triglyceride level is 500 mg/dl and over
* Significant abnormal liver dysfunction: AST, ALT level over or equal to 2.5 times, Total bilirubin level over or equal 2 times as high as upper normal limit(UNL)
* Significant abnormal renal dysfunction
* Anemia
* Abnormality of thyroid function(out of significant normal TSH range )
* Hepatitis B or C test is positive
* Pregnant women or nursing mothers
* Has a contraindication to treatment
* Fertile women who not practice contraception with appropriate methods
* Participated in other trial within 4 weeks
* Participating in other trial at present
* In investigator's judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin (HbA1c) | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from baseline in glycemic parameters | Baseline, 24 weeks
Change from baseline in HbA1c target achievement rate (HbA1c < 7%) | Baseline, 24 weeks
Change from baseline in lipid parameters | Baseline, 24 weeks
Evaluate safety of CKD-501 from physical exam, vital sign, laboratory test, adverse events | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SungWoo Park, M.D., Ph.D., Study Chair — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KS, Hong S, Ahn HY, Park CY. Comparative Efficacy of Lobeglitazone Versus Pioglitazone on Albuminuria in Patients with Type 2 Diabetes Mellitus. Diabetes Ther. 2021 Jan;12(1):171-181. doi: 10.1007/s13300-020-00948-1. Epub 2020 Oct 24. PMID 33099742